CLINICAL TRIAL: NCT04171882
Title: In Vivo Assessment of Neuroinflammation With 18-FDPA714 PET/CT
Brief Title: Microglial Cells Activation Imaging Using PET-CT With 18F-DPA714
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weibing Miao, PhD (Other)
Responsible Party: Sponsor-Investigator, Weibing Miao, PhD, professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA, ECFAH of FMU [2019]253
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Microglial Cells Activation Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is accumulating evidence suggesting that inflammatory processes, through microglial activation, would play a key role in brain injury and degeneration. It is considered that microglial activation would be part of self-propelling cycle of neuroinflammation that fuels Neurologic deterioration. It is however hard to evidence microglial activation in vivo: first, the investigators need very high-resolution imaging tools and then, the only ligand available to date, 11C-PK11195, has a low sensitivity and specificity and provided heterogeneous results. 18F-DPA-714 is a new PET ligand which labels microglial cells. The investigators aim to explore the clinical feasibility used PET-CT with 18F-DPA714 to monitor microglial cells activation of brain in several different disease. This study might reveal significant neuroinflammatory process in the brain. The results of this study might provide a new biomarker of disease pathological progression and help as identifying subjects who might most benefit from a specific anti-inflammatory drug.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Positron emission tomography scans were acquired more than twice
* Written informed consent was provided by the patients and their health care proxies -

Exclusion Criteria:

* Contraindication for PET examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with neurological or psychiatry diseases or known brain lesion
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Value (SUV) | 2 years
  Measures of specific binding of 18F-DPA-714 measures of specific binding of the tracer

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Miu weibing, Fuzhou
  - Yao shaobo, Tianjin